CLINICAL TRIAL: NCT00815204
Title: Measurement of Pituitary Volume and Hormonal Changes in Patients With Post-traumatic Stress Disorder
Status: Completed | Type: Observational
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Odelia Cooper, Odelia Cooper, MD, Cedars-Sinai Medical Center
Other Study IDs: 13353
Record Dates: First submitted 2008-12-24; First posted 2008-12-29 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Posttraumatic Stress Disorder
Keywords: PTSD; HPA axis; Pituitary volume
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Dexamethasone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Will be collecting blood to check for hormone levels
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- posttraumatic stress disorder
  Interventions: Procedure: MRI of the pituitary; Procedure: DEX/CRH test
- history of trauma exposure but no PTSD
  Interventions: Procedure: MRI of the pituitary; Procedure: DEX/CRH test
- healthy controls
  Interventions: Procedure: MRI of the pituitary; Procedure: DEX/CRH test

INTERVENTIONS:
Procedure: MRI of the pituitary — Patients will undergo a T1 weighted MRI of the pituitary to measure pituitary volume
  Other Names: MRI; Pituitary
Procedure: DEX/CRH test — Subjects will have blood drawn for baseline ACTH, cortisol, and other hormones and then undergo a DEX/CRH test. Will then measure ACTH and cortisol on test.
  Other Names: Dexamethasone; CRH

SUMMARY:
Approximately, post-traumatic stress disorder (PTSD) occurs in 8% of the adult population over time. Exposure to traumatic events increases the risk of poor physical health and often leads to disability. The biology of PTSD is continually being explored in order to help find better treatments for this debilitating disorder. In our study, we propose to further our understanding of PTSD. Prior research has found that patients with PTSD have changes in the stress hormone pathway. In this pathway, there is release of certain hormones from the pituitary gland in the brain that feed into the blood stream and tell the adrenal gland to produce stress hormones.

The pituitary is a gland located at the base of the brain which controls the hormones in the body, including the stress hormones. Research in other psychiatric disorders has found changes in the pituitary volume along with changes in the hormones. This has not been investigated yet in PTSD. Therefore, we propose in our study to measure pituitary volume in people with PTSD and look at the changes in the stress hormone pathway. Moreover, we will investigate whether other hormones are affected by PTSD. In this way, we can further our understanding of the the biology of PTSD and help develop new therapies which can intervene through the hormonal system.

DETAILED DESCRIPTION:
Lifetime prevalence of post-traumatic stress disorder (PTSD) is estimated at 8%. Exposure to traumatic events increases the risk of poor physical health, and chronic PTSD often leads to disability. The pathophysiology of PTSD is continually being explored in order to help find better treatment modalities for this debilitating disorder. Proposed mechanisms for the altered stress axis in PTSD include changes at the level of the pituitary. Though the pituitary stress hormone axis has been explored, no work has been done to evaluate for changes in the pituitary volume in response to these changes in the stress axis in PTSD. We have designed a study which will assess for differences in pituitary volumes. We will compare volumes in patients with PTSD, non-PTSD subjects who have had a history of trauma, and healthy controls. We will test the HPA axis through the dexamethasone/CRH test, a standardized diagnostic test, and correlate the findings with changes in the pituitary volume. Moreover, we will assess for changes in other endocrine axes and proteins.

We propose to further our understanding of PTSD by establishing a direct link between structure and function. By establishing these links in structure and function, novel therapies which can intervene through the endocrine system may prove to be of benefit in treating PTSD

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* history of PTSD

Exclusion Criteria:

* Uncontrolled medical or psychiatric conditions Liver or kidney disease Use of anti-depressants or ketoconazole Use of steroids within a year of the study Use of drugs of abuse Pregnancy or nursing Metal implants Low testosterone states A history of head bleeds or pituitary tumors

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects will be recruited from psychiatric clinics at Cedars-Sinai and at the West Los Angeles VA Center
Sampling Method: Non-Probability Sample
Enrollment: 39 (Actual)
Dates: Start 2008-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Pituitary volume | On second day of study

SECONDARY OUTCOMES:
Cortisol and ACTH levels on DEX/CRH test | On day 1 and day 2 of study test

CONTACTS AND LOCATIONS:
Overall Officials: Shlomo Melmed, MD, Study Director — Cedars-Sinai Medical Center; Odelia Cooper, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States